CLINICAL TRIAL: NCT03196661
Title: Preliminary Study on Safety and Immunogenicity of Influenza A (H7N9) Vaccine in the Population
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hualan Biological Bacterin Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2015L00054
Record Dates: First submitted 2017-05-19; First posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-05

CONDITIONS: Influenza A
Keywords: safety investigation

STUDY DESIGN:
Intervention Model Description: Subjects were inoculated with influenza A (H7N9) virus inactivated vaccine/split influenza vaccine or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial achieved the goal of random and blind method through blinded method for vaccine. All the testing vaccines and reference vaccines are provided by sponsor, and entrust Medical statistics unit to blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- H7N9 split influenza vaccine (15μg/dose) (Placebo Comparator): This group was divided into three subgroups according ages of subjects, the ages of those subjects are: 3 to 11(36 subjects got inoculated test vaccines, 18 subjects got inoculated reference vaccines)，12 to 17(36 subjects got inoculated test vaccines, 12 subjects got inoculated reference vaccines)，≥18 (36 subjects got inoculated test vaccines, 12 subjects got inoculated reference vaccines).
  Immune procedure: 0,21st day; Physical examination: 0,4th, 21st,25th day; Antibody detection: 0,21st,42nd day.
  Interventions: Biological: Influenza A (H7N9) virus vaccine
- H7N9 split influenza vaccine (30μg/dose) (Placebo Comparator): This group was divided into three subgroups according ages of subjects, the ages of those subjects are: 3 to 11(36 subjects got inoculated test vaccines, 18 subjects got inoculated reference vaccines)，12 to 17(36 subjects got inoculated test vaccines, 12 subjects got inoculated reference vaccines)，≥18 (36 subjects got inoculated test vaccines, 12 subjects got inoculated reference vaccines).
  Immune procedure: 0,21st day; Physical examination: 0,4th, 21st,25th day; Antibody detection: 0,21st,42nd day.
  Interventions: Biological: Influenza A (H7N9) virus vaccine
- H7N9 whole virus influenza vaccine (7.5μg/dose) (Placebo Comparator): This group was divided into two subgroups according ages of subjects, the ages of those subjects are: 12 to 17(54 subjects got inoculated test vaccines,18 subjects got inoculated reference vaccines)，≥18 (54 subjects got inoculated test vaccines, 18 subjects got inoculated reference vaccines).
  Immune procedure: 0,21st day; Physical examination: 0,4th, 21st,25th day; Antibody detection: 0,21st,42nd day.
  Interventions: Biological: Influenza A (H7N9) virus vaccine
- H7N9 whole virus influenza vaccine (15μg/dose) (Placebo Comparator): This group was divided into two subgroups according ages of subjects, the ages of those subjects are: 12 to 17(54 subjects got inoculated test vaccines,18 subjects got inoculated reference vaccines)，≥18 (54 subjects got inoculated test vaccines, 18 subjects got inoculated reference vaccines).
  Immune procedure: 0,21st day; Physical examination: 0,4th, 21st,25th day; Antibody detection: 0,21st,42nd day.
  Interventions: Biological: Influenza A (H7N9) virus vaccine

INTERVENTIONS:
Biological: Influenza A (H7N9) virus vaccine — To prevent the infection of H7N9 virus.

SUMMARY:
Adopt the design of random, blind method and placebo to parallel control and progressive methods of groups to study and evaluate the safety and immunogenicity of influenza A (H7N9) vaccine (two types, one type with two specifications) on people of different ages. The vaccines used for testing include: influenza A (H7N9) virus inactivated vaccine/split influenza vaccine (15μg /dose), influenza A (H7N9) virus inactivated vaccine/split influenza vaccine (30μg / dose), influenza A (H7N9) virus inactivated vaccine/whole influenza vaccine (7.5μg / dose) and influenza A (H7N9) virus inactivated vaccine/ whole influenza vaccine (15μg / dose).

The study between different subgroups was carried out in an orderly and progressive manner, that is, each kind of vaccine by the dose is from low to high according to the order of age from old to young. Firstly, the study on 15μg/dose split vaccine group (aged 18 and above) and 7.5μg/dose whole-virus vaccine group (aged 18 and above) was carried out and then the study on 15μg/dose split vaccine group (aged 12-17) and 7.5μg/dose whole-virus vaccine group (aged 12-17) was conducted upon 7-day safety was confirmed after the vaccination, finally the study on 30μg/dose split vaccine group (aged 18 and above) and 15μg/dose whole-virus vaccine group (aged 18 and above) was done. By that analogy for the same conditions, the next group of test can be done after the 7-day safety of the last group of vaccine is confirmed.

Subjects and researchers didn't know the formulations of the vaccines used. The vaccine is injected into the upper arm deltoid muscle. After 30 minutes of field observation on safety, the subjects' axillary temperature shall be recorded on the Record Book prepared by the research and local and systemic reactions to injection at the 6th, 24th, 48th, and 72th hour and on the 4th, 8th, 21st and 30th day shall also be recorded. This paper collected 5 serum samples: day 0 (before the first-dose vaccination), day 4 (after the first-dose vaccination), day 21 (before the second-dose vaccination), day 25 (fourth day after the second-dose vaccination) and day 42 (21st day after the second-dose vaccination), of which, blood samples on day 0, 21 and 42 should be stored at 18℃ for antibody detection and the remaining 2 blood samples are only used for blood routine examination, routine urine test, blood biochemistry and other laboratory examinations.

ELIGIBILITY:
Inclusion Criteria:

* Permanent healthy residents with normal intelligence meet the minimum age requirement. Literate and willing to provide written informed consent.
* A signed informed consent.
* Willing to comply with the rules of the clinical trial scheme. Accept the blood examination before and after immunization and cooperate follow-up visit.

Exclusion Criteria:

* Exclusion criteria of the first vaccination A person with a history of H7N9 virus infection or suspected infection; Who is allergic to any component of trial vaccine (and past history of any allergy vaccination), especially allergic to eggs; No spleen, or the spleen isn't working; Autoimmune diseases or immunodeficiency, have been treated with immunosuppressant over the past six months; Acute attack of acute illness or chronic disease in almost 7 days; Accept blood products in three months before getting inoculated testing vaccine; Got inoculated active virus vaccine in 14 days or subtype or inactivated virus in 7 days before getting inoculated testing vaccine; Who had been infected by any acute diseases ;
* Who had fever in past 3 days (axillary temperature ≥ 38 ℃);
* Who is participating another clinical trial
* Who had allergies, convulsions, epilepsy, encephalopathy, psychosis history or family history;
* Who is suffering from thrombocytopenia or other coagulation disorder, which may result to intramuscular injection contraindication; The laboratory detection indexes are abnormal before getting inoculated testing vaccine; The females are in suckling period, pregnancy, plan of pregnant or pregnancy tests (positive).
* Who had fever in the past 3 days (axillary temperature ≥ 37.1 ℃). Any other situations investigator think about may affect trial evaluation. Exclusion criteria of the second vaccination Level 3 and above allergic reactions (local and general side effect, vital signs and abnormal laboratory index) related to vaccine were appeared after the first vaccination.

Level 2 and above allergic reactions related to vaccine were appeared after the first vaccination.

-Any other situations investigator think about may affect trial evaluation.

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 588 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2016-07-05 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
587 subjects accept the observation of local adverse reaction according to Guidelines for grading standard of adverse reaction of clinical trial of vaccine used for prevention. | 20 days after the inoculation of first needle
  Inspect the measures like pain, induration, redness, red and swollen, rash, pruritus, skin mucosa reaction, etc. All these data is collected through questionnaires.
587 subjects accept the observation of local adverse reaction according to Guidelines for grading standard of adverse reaction of clinical trial of vaccine used for prevention. | 30 days after the inoculation of second needle
  Inspect the measures like pain, induration, redness, red and swollen, rash, pruritus, skin mucosa reaction, etc. All these data is collected through questionnaires.
587 subjects accept the observation of systemic adverse reactions according to Guidelines for grading standard of adverse reaction of clinical trial of vaccine used for prevention. | 20 days after the inoculation of first needle
  Inspect the measures like fever, headache, fatigue, weak, nausea, diarrhea, cough, allergic reaction, etc. All these data is collected through questionnaires.
587 subjects accept the observation of systemic adverse reactions according to Guidelines for grading standard of adverse reaction of clinical trial of vaccine used for prevention. | 30 days after the inoculation of second needle
  Inspect the measures like fever, headache, fatigue, weak, nausea, diarrhea, cough, allergic reaction, etc. All these data is collected through questionnaires.

SECONDARY OUTCOMES:
558 subjects accept the immunogenicity test according to micro-hemagglutination-inhibition test. | 21 days after the inoculation of first needle
  China pharmaceutical biological products analysis institute tests the HI antibody titer of H7N9 influenza virus in blood samples by adopting internationally-used micro-hemagglutination-inhibition test.
558 subjects accept the immunogenicity test according to micro-hemagglutination-inhibition test. | 42 days after the inoculation of second needle
  China pharmaceutical biological products analysis institute tests the HI antibody titer of H7N9 influenza virus in blood samples by adopting internationally-used micro-hemagglutination-inhibition test.